## Efficacy of near-assisted learning (NAL) in improving students' OSCE grades: A single-blinded RCT

Document date: 10/4/2019

## **Study protocol:**

In this single-blinded randomized controlled trial, 1<sup>st</sup> year male medical students of Sulaiman Alrajhi Colleges were invited via emails to participate voluntarily. Forty-eight students agreed to join and, after informed consent, were randomly assigned to one of two groups; the near-assisted learning group (The intervention) and the self-directed learning group (The control arm). Meanwhile, a group of 5<sup>th</sup> year medical students, known to be the top in their class, were invited to participate as instructors during the OSCE sessions. After their acceptance, they underwent extensive 2-week crash course focusing in basics of medical education, teaching and feedback cycle, along with quick supervised revision of systemic and general physical examination. At the analysis phase, scores of the previous batch were also included as a 3<sup>rd</sup> group for comparison. The study was concluded after 9 days, when the students had their skills evaluated during OSCE examination.

## Analysis plan:

Through SPSS 23<sup>rd</sup> edition, frequency, proportion analysis, chi-square and Fisher's exact test were used. A probability value of less than .05 was determined for significance.

## **Results:**

Those scoring B or better in the near-assisted learning, self-directed learning and the students of the previous batch groups were 22 (88%), 19 (82.6%) and 7 (50%), respectively (p= 0.025). More participants from the last group score A or more in comparison to the other two groups. On the other hand, less students failed the OSCE exam from the near-assisted and self-directed learning groups than the group of the prior batch.